CLINICAL TRIAL: NCT05762796
Title: Assessing the Efficacy of Alterations in Subcortical-Cortical Functional Connectivity From Transcranial Direct Current Stimulation in Older Children After Mild Traumatic Brain Injury
Brief Title: Neuromodulation and Neuroimaging in Older Children With Mild Traumatic Brain Injury
Acronym: CI-tDCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Ghazala Tanveer Saleem, Assistant Professor, State University of New York at Buffalo
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00006696; UL1TR001412 (NIH)
Record Dates: First submitted 2023-02-14; First posted 2023-03-10 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Brain Concussion; Mild Traumatic Brain Injury; Motor Disorders; Cognitive Impairment
Keywords: Brain Concussion; Mild Traumatic Brain Injury; Child; Motor Activity; Cognitive Impairment; Transcranial Direct Current Stimulation; Neuroimaging
MeSH Terms: conditions — Brain Concussion; Motor Disorders; Cognitive Dysfunction; Motor Activity | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: The Aim 1 of the study uses a cross-sectional design. The behavioral and neuroimaging data will be collected in one or two separate visits.
  The Aim 2 & Aim 3 of the study use a cross-over design. The data will be collected in either twenty-three or twenty-four visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Healthy Controls (No Intervention): Never-concussed age-and gender-matched healthy controls will not receive any intervention. Behavioral and neuroimaging measurements will be administered only once, at the initial visit.
- tDCS in Youth with mild traumatic brain injury (Experimental): Behavioral as well as neuroimaging measurements will be administered at the final post-anodal transcranial direct current stimulation (tDCS), final post-sham tDCS, and at 30-day follow-up visits.
  tDCS will be administered after the initial behavioral and neuroimaging testing. Ten sessions of 1.5 mA real tDCS and 10 sessions of sham tDCS will be administered using Neurocom (Germany) DC stimulator and two 5x7 electrodes, moistened in saline solution, to 10 participants with mTBI following a cross-over design with a 2-week washout period. The location of the brain regions will be determined using either the Transcranial Magnetic Stimulation Neuronavigation or Brainsight Neuronavigation system. The anode will be placed over pre-determined brain regions, whereas the cathode will be placed either over Fp2 (contralateral supraorbital) or other suitable reference areas.
  Interventions: Device: tDCS in Youth with mild traumatic brain injury

INTERVENTIONS:
Device: tDCS in Youth with mild traumatic brain injury — The safety and tolerability of tDCS have been established in children with mTBI (1). A recent study of 13-18 year youths post-mTBI showed that three sessions of 1.5 mA anodal tDCS over the left DLPFC, positively influenced prolonged working memory deficits. (2) Additionally, rodent studies show the effectiveness of tDCS in improving cognitive-motor (motor planning and balance/gait) function in rats with mTBI. (3)
  Arms: tDCS in Youth with mild traumatic brain injury

SUMMARY:
Mild traumatic brain injury (mTBI) often causes persistent motor and cognitive deficits in children resulting in functional limitations. We are testing a brain stimulation method along with evaluating objective tools to help record and restore communication among affected brain areas, which will facilitate recovery in youth after mTBI.

DETAILED DESCRIPTION:
About 1.9 million children sustain mTBI per year from sports injuries alone in the US. In about 30% of children, the cognitive-motor effects of mTBI interrupt typical neurodevelopment leading to chronic neurological conditions. The limited evidence available on mTBI suggests that residual symptoms may involve the brain stem (BS); the subcortical region that is now shown to influence cognitive-motor control. The BS also has functional interconnections to other cortical regions involved in cognitive-motor learning such as the dorsolateral prefrontal cortex, premotor cortex, and primary motor cortex. While clinicians examine certain risk factors such as amnesia and history of prior concussions, they lack objective biomarkers to accurately predict the post-mTBI prognosis in children, and to accurately guide treatment. Further, there is no evidence-based standard of care established, so children may be released to pre-injury activity levels before full neurophysiological recovery, predisposing them to further mTBI and associated sequelae.

Transcranial Direct Current Stimulation (tDCS), a non-invasive treatment, has been demonstrated to positively influence cognitive-motor control by modulating the excitability of both cortical and subcortical structures. Additionally, resting state functional connectivity has shown promise in diagnosing and predicting recovery in adult TBI. However, the efficacy of tDCS for children with mTBI is not yet established due to their atypical cortical activity and variable symptomology. Consequently, we aim to determine the efficacy of tDCS for promoting recovery in 10 youths (aged 10 to 15 years) who exhibit persistent symptoms of mTBI using a cross-over design compared with 10 never-injured youths as controls, and to test the application of neural correlates to provide insights into their functional change and recovery by comparing group differences.

ELIGIBILITY:
Experimental Cohort:

Inclusion Criteria:

* age 10-15 years at enrollment
* enrolled after 6 weeks of mTBI injury
* exhibiting post-concussive symptoms (e.g., difficulty planning, sequencing, and executing a motor action)
* Sustained an mTBI or concussion within the past 12 months
* Parent and child proficient in English

Healthy Controls Cohort:

Inclusion Criteria:

* 10 to 15 years old
* no concussion history
* Parent and child proficient in English

Experimental Cohort:

Exclusion Criteria:

* loss of consciousness > 30 minutes
* post-traumatic amnesia > 24 hours
* intracranial findings on clinical imaging
* history of developmental delay
* history of learning disability or ADHD
* Sustained a lower limb or upper limb injury that has not healed
* History of Seizures
* Noticeable skin lesions/burns or any other severe skin problems at the site of the electrodes before the start of the stimulation.
* Parent/guardian report metal implants anywhere in the head/ncek/body on the MRI screening form (see attached).
* Parent/guardian report shrapnel/bullets in the body on the MRI screening form.
* Parent/guardian report any electronic implant such as a cardiac pacemaker, cochlear implant, ventricular shunt, cardiac defibrillator, aneurysm clips, pacing wires, any implant held in place with a magnet, heart valve, or deep brain stimulator on the MRI screening form.
* Parent/guardian report a craniotomy or any other surgery in the past 6 weeks on the MRI screening form.
* Parent/guardian report being claustrophobic on the MRI screening form.
* Parent/guardian report and provide orbit x-ray after the eye injury involving a metal that the subject is cleared as indicated on the MRI screening form.
* Pregnant females as reported by parent/guardian on the pre-consent screening form. Pubertal/post-pubertal female participants14 and above will be provided a separate post-consent screening form at each MRI visit to ensure the female reports accurately without fear.

Healthy Controls Cohort:

Exclusion Criteria:

* diagnosed with developmental delay
* sustained a lower limb or upper limb injury that has not healed
* history of Learning Disability and/or ADHD
* Parent/guardian report metal implants anywhere in the head/ncek/body on the MRI screening form (see attached).
* Parent/guardian report shrapnel/bullets in the body on the MRI screening form.
* Parent/guardian report any electronic implant such as a cardiac pacemaker, cochlear implant, ventricular shunt, cardiac defibrillator, aneurysm clips, pacing wires, any implant held in place with a magnet, heart valve, or deep brain stimulator on the MRI screening form.
* Parent/guardian report a craniotomy or any other surgery in the past 6 weeks on the MRI screening form.
* Parent/guardian report being claustrophobic on the MRI screening form.
* Parent/guardian report and provide orbit x-ray after the eye injury involving a metal that the subject is cleared as indicated on the MRI screening form.
* Pregnant females as reported by parent/guardian on the pre-consent screening form. Post-pubertal females 14 and above will be provided a separate post-consent screening form at each MRI visit to ensure the female reports accurately without fear.

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Changes in the Revised Physical and Neurological Examination of Subtle Signs (PANESS - Gaits and Stations Measures) | Day 1 (at the initial visit), Day 26- 30 (final post-anodal transcranial direct current stimulation (tDCS), Day 60 -64 (final post-sham tDCS), and Day 94 (at 30-days follow up visit).
  The PANESS is used to assess static and dynamic postural stability of adolescents. The PANESS contains nine static and dynamic balance tasks: 1) walking on heels, 2) walking on toes, 3) walking on sides of feet, 4) double-legged stance, 5) single-legged stance for 30 seconds, 6) tandems stance for 20 seconds, 7) forward tandem walking, 8) backward tandem walking, and 9) hopping in place on one foot. The scores from all tasks are combined to form an aggregated score.
Changes in the Nine-Hole Peg Test | Day 1 (at the initial visit), Day 26- 30 (final post-anodal transcranial direct current stimulation (tDCS), Day 60 -64 (final post-sham tDCS), and Day 94 (at 30-days follow up visit).
  The test consists of a square board with 9 holes. The participants are asked to pick up pegs one at a time and place them into holes as quickly as possible. The participants are then instructed to remove the pegs one by one from the board and put them back into the container. The average time from four trials is examined to arrive at the total score.
Changes in the Dual-Task Screen | Day 1 (at the initial visit), Day 26- 30 (final post-anodal transcranial direct current stimulation (tDCS), Day 60 -64 (final post-sham tDCS), and Day 94 (at 30-days follow up visit).
  It consists of a gait task and an eye-hand coordination task. In the single gait task condition, participants are instructed to walk as quickly as possibly for 6 meter and step over a 1.5 meter obstacle placed 4 meter from the start. In the dual gait condition, participants will repeat the gait task while counting the months of the year backward. In the eye-hand coordination single task, participants will be instructed to stand 1.5 meter away from the wall and throw and catch a tennis ball for 30 seconds. In the dual task eye-hand coordination condition, the participants will repeat the catch and throw task while serially subtracting 3s from 100s. The difference between the single task and the dual task will be calculated to arrive at the score for each participant.
Changes in Motor Control Test Measurements (Posturography) | Day 1 (at the initial visit), Day 26- 30 (final post-anodal transcranial direct current stimulation (tDCS), Day 60 -64 (final post-sham tDCS), and Day 94 (at 30-days follow up visit).
  The motor control test (MCT) will be administered using the Posturography Machine to assess the ability of the patient to recover from translational disturbances of the support surface. The six conditions each participant will perform include three forward translations with small, medium, and large intensities as well as three backward translations with small, medium, and large intensities. Each participant go through three trials at each translation and intensity. The participant will be scored on latency; their ability to respond to the translation in milliseconds, and the amplitude scaling; the average amount of weight carried by each leg during the translation. An increased latency indicates impairment within the neural pathways that cause musculoskeletal problems in addition to central abnormalities. Abnormal amplitude scaling indicates inadequate or asymmetrical level of force exerted during the recovery from the support disturbance.
Changes in resting-state functional magnetic resonance imaging outcome | Day 2-5 (post initial behavioral testing), Day 26- 32 (final post-anodal transcranial direct current stimulation (tDCS), Day 60 -66 (final post-sham tDCS), and Day 94 - 96 (post 30-days follow up behavioral testing visit).
  MRI scanning will be used to assess the functional connectivity among the brain areas involved in motor learning and motor planning. Functional connectivity will be measured by looking at differences in the control group and the experimental group.

SECONDARY OUTCOMES:
Changes in PHQ-8 | Day 1 (at the initial visit), Day 26- 30 (final post-anodal transcranial direct current stimulation (tDCS), Day 60 -64 (final post-sham tDCS), and Day 94 (at 30-days follow up visit).
  This 8-item questionnaire assesses depression in children. The scores of all variables will be aggregated to form a total score.
Changes in GAD-7 | Day 1 (at the initial visit), Day 26- 30 (final post-anodal transcranial direct current stimulation (tDCS), Day 60 -64 (final post-sham tDCS), and Day 94 (at 30-days follow up visit).
  This 7-item questionnaire assesses anxiety in children. The scores of all variables will be aggregated to form a total score.
Changes in WASI-II | Day 1 (at the initial visit), Day 26- 30 (final post-anodal transcranial direct current stimulation (tDCS), Day 60 -64 (final post-sham tDCS), and Day 94 (at 30-days follow up visit).
  This measure assesses overall cognitive abilities in children. The scores of all variables will be aggregated to form a total score.

CONTACTS AND LOCATIONS:
Overall Officials: Ghazala Saleem, EdD, Principal Investigator — State University of New York at Buffalo
Locations (1):
- Ghazala Saleem, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
MRI data is de-identified and available to Center for Brain Imaging (CBI) personnel and a limited number of CBI users who have signed authorized access agreements. CBI personnel and users will make a request in writing to PI and CBI study team member (Dr. Schweser) regarding the data release indicating the purpose for data use. To minimize risks to participants' privacy, a committee of experts will carefully review every data request from other scientists before allowing them to use this controlled-access database, to make sure they can also protect participants'' personal information. These other investigators may be at an institute of the Buffalo Translational Consortium or other research centers (academic or commercial) around the world
Supporting Information: Study Protocol
Time Frame: MRI data will become available after the study is finished. Data will be available indefinitely.
Access Criteria: Data can be accessed through Center for Brain Imaging database after written approval.

REFERENCES:
- [Background] Saleem GT, Crasta JE, Slomine BS, Cantarero GL, Suskauer SJ. Transcranial Direct Current Stimulation in Pediatric Motor Disorders: A Systematic Review and Meta-analysis. Arch Phys Med Rehabil. 2019 Apr;100(4):724-738. doi: 10.1016/j.apmr.2018.10.011. Epub 2018 Nov 7. PMID 30414398
- [Background] Brunoni AR, Amadera J, Berbel B, Volz MS, Rizzerio BG, Fregni F. A systematic review on reporting and assessment of adverse effects associated with transcranial direct current stimulation. Int J Neuropsychopharmacol. 2011 Sep;14(8):1133-45. doi: 10.1017/S1461145710001690. Epub 2011 Feb 15. PMID 21320389
- [Background] Rotter J, Kamat D. Concussion in Children. Pediatr Ann. 2019 Apr 1;48(4):e182-e185. doi: 10.3928/19382359-20190326-01. PMID 30986320
- [Background] Fregni F, Nitsche MA, Loo CK, Brunoni AR, Marangolo P, Leite J, Carvalho S, Bolognini N, Caumo W, Paik NJ, Simis M, Ueda K, Ekhitari H, Luu P, Tucker DM, Tyler WJ, Brunelin J, Datta A, Juan CH, Venkatasubramanian G, Boggio PS, Bikson M. Regulatory Considerations for the Clinical and Research Use of Transcranial Direct Current Stimulation (tDCS): review and recommendations from an expert panel. Clin Res Regul Aff. 2015 Mar 1;32(1):22-35. doi: 10.3109/10601333.2015.980944. PMID 25983531